CLINICAL TRIAL: NCT02011620
Title: Influence of Nitrates on Bone Remodeling and Endothelial Function in Patients With Type 2 Diabetes Mellitus.
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The sponsor was no longer in a position to sponsor a CTIMP. Study did not open.
Sponsor: Tameside Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Edward Jude, Consultant Diabetologist and Endocrinologist, Tameside Hospital NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D001
Record Dates: First submitted 2013-11-26; First posted 2013-12-13 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Endothelial Dysfunction; Bone Disease
MeSH Terms: conditions — Bone Diseases | interventions — isosorbide-5-mononitrate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Isosorbide-5-mononitrate (Active Comparator): Tablet Isosorbide mononitrate 20 mg; 1 tablet to be taken daily at night for a total duration of 6 months.
  Interventions: Other: Isosorbide-5-mononitrate
- Standard care (No Intervention): Standard care - no intervention with nitrates

INTERVENTIONS:
Other: Isosorbide-5-mononitrate — Tablet Isosorbide mononitrate 20 mg; 1 tablet to be taken daily at night for a total duration of 6 months.
  Other Names: Name of the MA holder: TEVA UK LIMITED; MA number (if MA granted by a Member State): PL 0289/0287; UNITED KINGDOM
  Arms: Isosorbide-5-mononitrate

SUMMARY:
Type 2 diabetes mellitus (DM) is becoming a leading global epidemic. DM affects several systems in the body. Most of the complications encountered in DM are attributed to uncontrolled hyperglycemia or poor glycemic control. Hyperglycemic stress tends to damage the inner lining of the small blood vessels (endothelium). Normally, the endothelium releases a chemical substance called nitric oxide (NO) which relaxes the blood vessels and also prevents blockade of these vessels. Therefore damage to the endothelium (endothelial dysfunction) results in diminished levels of NO which ultimately leads to occlusion of these small blood vessels (microvascular occlusion). Microvascular occlusion of vessels supplying the eyes, kidneys and nerves leads to serious complications like diabetic retinopathy, nephropathy and neuropathy.

Of late, the skeletal system has emerged as another vulnerable target of diabetic microvascular disease. Patients with DM have an increased risk of developing fractures. Certain predisposing factors like diabetic neuropathy and visual disturbances (retinopathy and cataract) increases the likelihood of fractures in DM. More recently, evolving research has demonstrated NO's prospective role in bone preservation. Earlier studies have also validated the use of nitrates (donor of NO) in improving bone strength and reducing the risk of fractures.

So far no study has investigated the effect of nitrates on endothelial function and bone microarchitecture in patients with diabetes. The investigators therefore propose to investigate the influence of nitrates on endothelial dysfunction and bone integrity in patients with type 2 diabetes. 40 patients with type 2 DM will be recruited into the study; 20 patients will receive 20 mg of oral isosorbide mononitrate daily and the other 20 will not receive the study drug. The investigators hope to demonstrate an improvement in endothelial function (by measuring skin blood flow) and bone integrity (by measuring markers of bone formation and bone resorption and bone mineral density - BMD) following 6 months of nitrate therapy.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is a chronic debilitating disease that affects almost all the systems in the body with accompanying diabetic complications (neuropathy, retinopathy and nephropathy) adding to the global burden of DM. These diabetic complications arise as a manifestation of hyperglycaemic damage induced at the cellular level particularly the endothelial cells (EC). Exposure to hyperglycaemic stress causes endothelial dysfunction, which is the major perpetrator of microvascular disease. Disruption of endothelial function also marks the advent of the subsequent development of cardiovascular disease (CVD) that includes atherosclerosis and coronary artery disease (CAD). Microvascular disease occurs as a result of deficiency of a potent endothelial vasodilator, nitric oxide (NO). NO plays a fundamental role in vascular regulation which is mediated through vasodilation. Other favourable characteristics of NO include antiplatelet activity and prevention of vascular smooth muscle cell (VSMC) proliferation. Unsurprisingly, diminished NO levels in DM will eventually lead to occlusion of the microvasculature in the retina, glomerulus and peripheral nerve (vasa nervorum).

Of late, the skeletal system has also emerged as another vulnerable target of diabetic microvascular disease. Certain predisposing factors like diabetic neuropathy (DN), visual disturbances (retinopathy and cataract), gait abnormalities and hypoglycemia increase the likelihood of fractures in DM. Among these factors DN contributes to a major extent in the development of fractures especially fractures of the lower extremities.

Current antiresorptive therapies include estrogen/ HRT (Hormone replacement therapy), bisphosphonates (BPP), selective estrogen receptor modulators (SERM) and denosumab (DMB). These agents mainly retard bone resorption in the trabecular bone, with minimal effects on cortical bone and are associated with only a 20-30% reduction in the risk of non-vertebral fractures. Moreover, they decrease bone formation and are not devoid of adverse effects. Some of these agents are also expensive and at times unavailable in some countries. All these limitations challenge the discovery of an ideal agent that can prevent bone resorption, increase bone formation and also reduce the risk of non-vertebral fractures.

Lately the therapeutic role of organic nitrates (source of NO) in bone metabolism has led to a breakthrough in this field of research. Nitrates are commonly used in the treatment of angina. Since nitrates are widely available, inexpensive and associated with limited side effects, it would be practical to exploit these characteristic features in the treatment of bone disease and endothelial dysfunction in DM.

AIMS

This pilot study aims to investigate the effect of Isosorbide mononitrate in patients with type 2 DM with respect to:

* Its influence on bone remodelling by assessing the levels of bone markers and its ability to improve BMD.
* Its role in modulating endothelial dysfunction.

HYPOTHESIS

In this randomised pilot study, patients with type 2 DM who receive 20 mg of Isosorbide mononitrate will show:

* An improvement in bone formation as measured by serum procollagen type 1 amino terminal propeptide (P1NP)
* Suppression of bone resorption as assessed by measurement of serum C-terminal cross-linked telopeptide of type-I collagen (CTX)
* Improvement in calcaneal BMD
* Improvement in endothelial mediated vasodilation.

PATIENTS 40 female/ male subjects with type 2 DM will be considered eligible for the study. They will be recruited from the Tameside Diabetes Centre and appropriate GP practices and a written consent will be obtained from them prior to participation in the study.

Since there is no placebo in this study, the research fellow and research nurse will be blinded to the treatment the patient is receiving. As it is known that the duration of diabetes can affect microvascular circulation and possibly bone metabolism, the two groups will be matched for the following variables: age, gender, duration of diabetes and severity of neuropathy.

Diabetes self-education and management along with dietary advice will be provided to all the participants in the study.

RANDOMISATION

With the help of a computer-generated program the study participants will be randomised into 2 groups:

* Group 1: 20 subjects will receive 20 mg/day of isosorbide mononitrate orally
* Group 2: 20 subjects will receive standard care

MEASUREMENTS Biochemical parameters at baseline and 6 months later

* Serum procollagen type 1 amino terminal propeptide (P1NP), a marker of bone formation which indicates osteoblastic activity.
* Serum C-terminal cross-linked telopeptide of type-I collagen (CTX), a marker of bone resorption Clinical parameters at baseline
* Laser Doppler imaging
* Calcaneal BMD (Sahara clinical bone sonometer; Hologic, Waltham, MA) Blood samples will be obtained from the antecubital vein following an overnight fast and after resting for 15 minutes in the supine position.

Assessment of the microcirculation with Laser Doppler Iontophoresis at baseline and 6 months A standard measurement of microcirculation is laser Doppler iontophoresis, which is used by several research institutes. In this trial the skin microcirculation will be measured on the ventral aspect of the forearm using a Perimed Laser Doppler imager and iontophoresis system.

Endothelial-mediated vasodilation will be measured by the iontophoresis of acetylcholine, while sodium nitroprusside will be used to measure endothelium-independent vasodilation. The iontophoresis system consists of an ION chamber (iontophoresis delivery vehicle device) that sticks firmly to the skin and a reference electrode. The response in blood flow will be imaged and quantified using the Perimed Laser Doppler Imager (Sweden).

Assessment of calcaneal BMD at baseline and at 6 months This is a simple and convenient method to assess peripheral BMD and assess fracture risk. The device used is a quantitative ultrasound called Sahara Clinical Bone Sonometer (Sahara Clinical Bone Sonometer; Hologic, Waltham, MA). The calcaneus is the preferred peripheral site to assess fracture risk. This device uses ultrasound waves to determine the BMD of the calcaneus. In this procedure, once the bare heel is placed in the device, the BMD is calculated within 30 seconds and the results are then generated on paper by the device.

STATISTICAL ANALYSIS The results obtained from this study will be reported as a difference between the baseline and 6 months later following a single daily oral dose of 20 mg isosorbide mononitrate. The difference between the 2 groups will also be inferred at the end of 6 months. The changes in skeletal parameters (serum P1NP and CTX) and microcirculation will be compared between the 2 groups using t-tests to determine post hoc differences. A p-value of < 0.05 will be considered significant. All analyses will be conducted using the Statistical Package for Social Sciences (SPSS Inc., Chicago, Illinois, USA).

DURATION OF THE STUDY The estimated time for enrolment of patients will be within 6 months. The duration of the study is 6 months and the last follow up will be at the end of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Females and males aged between 40-75 years
* A diagnosis of type 2 DM based on one of the following criteria (ADA - 2010):
* Fasting plasma glucose (FPG) >= 126 mg/dL (7.0 mmol/L) or
* 2-h plasma glucose >= 200 mg/dl (11.1 mmol/L) during an OGTT or
* Classic symptoms of hyperglycemia or hyperglycemic crisis with a random plasma glucose >= 200 mg/dL (11.1 mmol/L).
* Known history of type 2 diabetes mellitus on treatment

Exclusion Criteria:

* At screening, age below 40 years and above 75 years.
* Pregnancy or lactation
* Type 1 diabetes mellitus (patients with a history of ketoacidosis, age of onset of DM before 25 years of age, BMI <21 kg/m2 and use of insulin without a concomitant oral hypoglycemic agent)
* Patients with uncontrolled hypertension (systolic blood pressure [SBP] > 160/90 mmHg) or hypotension (SBP of <=100 mm Hg) at screening.
* History of hypersensitivity to nitrates
* History of low blood pressure
* History of raised intracranial pressure (from cerebral haemorrhage or head trauma)
* History of cardiovascular disease (ischaemic heart disease, previous stroke and severe peripheral vascular disease [Ankle brachial pressure index - ABPI< 0.7])
* History of acute circulatory failure (shock), circulatory collapse, cardiogenic shock
* History of hypertrophic obstructive cardiomyopathy, constrictive pericarditis, cardiac tamponade, low cardiac filling pressures, aortic/ mitral valve stenosis
* History of general systemic illness including cardiac, hepatic or renal insufficiency
* Patients with clinical nephropathy (24 hour protein > 0.5g or dipstix protein +) or renal failure (serum creatinine > 130 µmol/l).
* History of anaemia
* History of closed angle glaucoma
* History of migraine headaches
* History of hypothyroidism
* History of hypothermia
* History of malnutrition
* History of Paget's disease and other metabolic bone disorders
* History of coeliac or inflammatory bowel disease
* History of multiple myeloma or cancer
* History of nitrate use for cardiac conditions
* History of treatment with phosphodiesterase type-5 inhibitors
* History of foot ulcers
* History of active foot deformities e.g. Charcot foot
* History of glucocorticoid intake within the last 3 months
* History of hormone replacement therapy in the last 12 months
* History of treatment with SERM (selective estrogen receptor modulator)
* History of treatment with thiazolidinedione
* History of anticonvulsant use
* History of past or current treatment for osteoporosis
* History of bisphosphonate therapy within the last 3 years

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10 (Estimated); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Improvement in endothelial function as measured by laser doppler imaging. | 6 months
  Assessment of the microcirculation with Laser Doppler Iontophoresis at baseline and 6 months
  A standard measurement of microcirculation is laser Doppler iontophoresis, which is used by several research institutes. In this trial the skin microcirculation will be measured on the ventral aspect of the forearm using a Perimed Laser Doppler imager and iontophoresis system.
  Endothelial-mediated vasodilation will be measured by the iontophoresis of acetylcholine, while sodium nitroprusside will be used to measure endothelium-independent vasodilation. The iontophoresis system consists of an ION chamber (iontophoresis delivery vehicle device) that sticks firmly to the skin and a reference electrode. The response in blood flow will be imaged and quantified using the Perimed Laser Doppler Imager (Sweden).

SECONDARY OUTCOMES:
Improvement in bone metabolism | 6 months
  1. An improvement in bone formation as measured by serum procollagen type 1 amino terminal propeptide (P1NP)
  2. Suppression of bone resorption as assessed by measurement of serum C-terminal crosslinked telopeptide of type 1 collagen (CTX)
  3. Improvement in calcaneal bone mineral density

CONTACTS AND LOCATIONS:
Overall Officials: Edward Jude, MD, MRCP, Principal Investigator — Tameside General Hospital NHS Foundation Trust
Locations (1):
- Tameside General Hospital NHS Foundation Trust, Manchester, United Kingdom

REFERENCES:
- [Background] Wimalawansa SJ. Nitric oxide: new evidence for novel therapeutic indications. Expert Opin Pharmacother. 2008 Aug;9(11):1935-54. doi: 10.1517/14656566.9.11.1935. PMID 18627331
- [Background] Veves A, Akbari CM, Primavera J, Donaghue VM, Zacharoulis D, Chrzan JS, DeGirolami U, LoGerfo FW, Freeman R. Endothelial dysfunction and the expression of endothelial nitric oxide synthetase in diabetic neuropathy, vascular disease, and foot ulceration. Diabetes. 1998 Mar;47(3):457-63. doi: 10.2337/diabetes.47.3.457. PMID 9519754
- [Background] Mascarenhas JV, Jude EB. Pathogenesis and medical management of diabetic Charcot neuroarthropathy. Med Clin North Am. 2013 Sep;97(5):857-72. doi: 10.1016/j.mcna.2013.05.002. PMID 23992897
- [Background] Wimalawansa SJ. Rationale for using nitric oxide donor therapy for prevention of bone loss and treatment of osteoporosis in humans. Ann N Y Acad Sci. 2007 Nov;1117:283-97. doi: 10.1196/annals.1402.066. PMID 18056048
- [Background] Jamal SA, Cummings SR, Hawker GA. Isosorbide mononitrate increases bone formation and decreases bone resorption in postmenopausal women: a randomized trial. J Bone Miner Res. 2004 Sep;19(9):1512-7. doi: 10.1359/JBMR.040716. Epub 2004 Jul 26. PMID 15312252
- [Background] Jamal SA, Goltzman D, Hanley DA, Papaioannou A, Prior JC, Josse RG. Nitrate use and changes in bone mineral density: the Canadian Multicentre Osteoporosis Study. Osteoporos Int. 2009 May;20(5):737-44. doi: 10.1007/s00198-008-0727-7. Epub 2008 Sep 18. PMID 18800179 (Retraction: PMID 27909783 Osteoporos Int. 2016 Dec 1;:)